CLINICAL TRIAL: NCT02638116
Title: Open-Label, Sequential-Design Drug Interaction Study of the Effect of Omeprazole on the Pharmacokinetics of Ibrutinib in Healthy Adults
Brief Title: A Drug Interaction Study to Assess the Effect of Omeprazole on the Pharmacokinetics of Ibrutinib in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108106; 2015-005015-32 (EudraCT Number); PCI-32765CLL1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Ibrutinib; Proton pump inhibitors; Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — ibrutinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib + Omeprazole (Experimental): Participants will receive a dose of Ibrutinib 560 milligram (mg) orally (4 x 140 mg capsules) on Day 1 and Day 7 and Omeprazole at a dose of 40 mg tablets orally once on Days 3 through 7.
  Interventions: Drug: Ibrutinib; Drug: Omeprazole

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered at a dose of 560 milligram (mg) orally (4 x 140 mg capsules) on Day 1 and Day 7.
Drug: Omeprazole — Omeprazole will be administered at dose of 40 mg tablets orally once daily from Day 3 to Day 7.

SUMMARY:
The purpose of this study is to evaluate the Effect of Omeprazole on the Pharmacokinetics of Ibrutinib in Healthy Adults.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, sequential-design drug interaction study to assess the effect of omeprazole on pharmacokinetics of ibrutinib and metabolite PCI-45227 in healthy participants. The study mainly consists of 3 Phases: Screening Phase (within 21 days prior to the first dose of study medication), treatment Phase, and a follow up Phase (10 to 12 days after the last dose of study medication). In the treatment Phase, participants will receive Ibrutinib 560 milligram (mg) orally (4 x 140 mg capsules) on Day 1 and Day 7. participants will receive Omeprazole at a dose of 40 mg tablets orally once on Days 3 through 7. The total duration of study for each participant will be approximately for 29 to 32 days. Blood samples will be collected for evaluation of pharmacokinetics of Ibrutinib. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* If a woman, must not be of childbearing potential: postmenopausal ( greater than [>] 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) >40 International units [IU]/ Liter [L]); surgically sterile
* If a woman, must have a negative serum β-human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine pregnancy test on Day-1
* Willing to adhere to the prohibitions and restrictions specified in the protocol
* If a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 milliliter [mL]/ minute [min]), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry, at Screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled until completion of the study
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-IV) criteria within 2 years before Screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at Screening and Day-1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Ibrutinib | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The Cmax is the maximum observed plasma concentration of Ibrutinib.
Time to Reach the Maximum Plasma Concentration (Tmax) of Ibrutinib | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The Tmax is the time to reach the maximum observed plasma concentration of Ibrutinib.
Area Under the Plasma Concentration-Time Curve From 0 to 48 Hours (AUC[0-48]) Post Dose of Ibrutinib | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The AUC (0-48hrs) is the area under the plasma Ibrutinib concentration-time curve from 0 to 48 hours post dosing.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) of Ibrutinib | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The AUC (0-last) is the area under the plasma Ibrutinib concentration-time curve from time 0 to time of the last observed quantifiable concentration (C[last]).
Metabolite to Parent (M/P) Ratio of Ibrutinib | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  Ratio of ibrutinib metabolite concentration to parent compound (ibrutinib) concentration will be assessed.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of PCI-45227 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The Cmax is the maximum observed plasma concentration of PCI-45227.
Time to Reach the Maximum Plasma Concentration (Tmax) of PCI-45227 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The Tmax is the time to reach the maximum observed plasma concentration of PCI-45227.
Area Under the Plasma Concentration-Time Curve From 0 to 48 Hours (AUC[0-48]) Post Dose of PCI-45227 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The AUC (0-48hrs) is the area under the plasma PCI-45227 concentration-time curve from 0 to 48 hours post dosing.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) of PCI-45227 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose on Day 1 and Day 7
  The AUC (0-last) is the area under the plasma PCI-45227 concentration-time curve from time 0 to time of the last observed quantifiable concentration (C[last]).
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (10 plus [+] / minus [-] 2 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium

REFERENCES:
- [Derived] de Jong J, Haddish-Berhane N, Hellemans P, Jiao J, Sukbuntherng J, Ouellet D. The pH-altering agent omeprazole affects rate but not the extent of ibrutinib exposure. Cancer Chemother Pharmacol. 2018 Aug;82(2):299-308. doi: 10.1007/s00280-018-3613-9. Epub 2018 Jun 7. PMID 29882017